CLINICAL TRIAL: NCT04609943
Title: Safety and Tolerability of Adaptive Escalating Multiple Doses (Three Times Daily) of a Soluble Guanylate Cyclase (sGC) Activator Inhale, BAY 1211163, as Inhalation in Intubated and Mechanically Ventilated Adult Patients With Moderate and Severe Acute Respiratory Distress Syndrome (ARDS). A Pilot (Phase Ib), First in Patient, Open Label Study
Brief Title: Study to Find the Highest Safe Dose of Soluble Guanylate Cyclase (sGC) Activator, BAY 1211163 Administered as Multiple Doses by Inhalation to Patients Who Cannot Breathe by Their Own and Suffer From a Type of Lung Failure That Causes Fluid to Build up in the Lungs Making Breathing Difficult (ARDS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Decision.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20425; 2019-004950-26 (EudraCT Number)
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAY1211163 (Experimental): Adult patients with moderate or severe Acute Respiratory Distress Syndrome (ARDS) diagnosis before study inclusion will receive BAY1211163.
  Interventions: Drug: BAY1211163

INTERVENTIONS:
Drug: BAY1211163 — Participants will receive one of the drug doses of BAY1211163 solution three times per day (TID) by inhalation for seven days.

SUMMARY:
With this study researchers want to find the highest safe dose of the soluble Guanylate Cyclase (sGC) Activator, BAY 1211163 and how safe and well the study drug works. Furthermore researchers want to gather information on the way the body absorbs, distributes and gets rid of the study drug given as increasing multiple doses by inhalation to patients who cannot breathe by their own and suffer from a type of lung failure that causes fluid to build up in the lungs making breathing difficult (ARDS)

ELIGIBILITY:
Inclusion Criteria:

* Intubated, mechanically ventilated moderate or severe ARDS patients [diagnosed according to Berlin definition of ARDS, including PEEP ≥ 5 cmH2O, X-ray, with PaO2/FiO2 between 80 and 200 mmHg (inclusive).
* Initial diagnosis of ARDS prior to study inclusion, confirmation of ongoing moderate or severe ARDS with PaO2/FiO2 between 80 and 200 mmHg (inclusive) during this time under maintained invasive mechanical ventilation.
* Hypoxemia with PaO2/FiO2 between 80 and 200 mmHg (inclusive) maintained for at least 8 hours (recommend to be 12 hours) after screening, despite consent to follow recommendation on ventilator strategy and PEEP management.
* Time from intubation must be ≤ 96h.
* Male and non-pregnant female.
* Informed consent of capable patient or, in case of patient being incapable of giving informed consent, consent for study inclusion will be sought according to applicable laws and regulations.

Exclusion Criteria:

* PaO2/FiO2 > 200 mmHg or < 80 mmHg at time of evaluation for inclusion.
* Moribund participants not expected to survive 24 hours (clinical decision).
* Expected duration of invasive mechanical ventilation less than 96 hours (clinical decision).
* History of pneumectomy or lung transplant.
* Current lung malignancy (including lung metastasis), or other malignancy requiring chemotherapy or radiation within the last month.
* History of chronic kidney disease and requiring renal replacement therapy dialysis at screening and/or baseline.
* Chronic liver disease Child-Pugh Class B and C.
* Hypoalbuminemia - serum albumin < 2.0 g/dL.
* Acute left ventricular failure and/or Left Ventricular Ejection Fraction < 30 %.
* Severe bronchopulmonal fistula.
* Clinical suspicion of pulmonary veno-occlusive disease.
* Heart right-sided endocarditis, tumors or mass.
* Rescue procedures already initiated at screening and/or Day 1.
* Use of co-medications involving moderate and strong inhibitors for CYP2C8 liver enzymes one week before assignment to intervention or during intervention.
* Off-label use of medication to treat Coronavirus SARS-CoV-2 virus unless recommended by scientific guidelines and accepted by DMC, investigator and sponsor.
* Plan to participate or past participation (within 30 days prior to Study Day 1) in other interventional studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Numbers of participants with treatment emergent adverse events (TEAEs) | Up to 9 days
Numbers of participants with dose limiting events (DLEs) | Day 1 to 7 (may include Day 8)
  A dose limiting event is defined as any of the TEAEs occurring during dosing with BAY1211163 and regarded by the investigators to be related to BAY1211163.

SECONDARY OUTCOMES:
Values of oxygenation index (OI) | Up to 28 days
  The Oxygenation Index (OI) is calculated by using the fraction of inspired oxygen (FiO2), the partial pressure of oxygen in arterial blood (PaO2) and the mean airway pressure (MPAW)

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Universitätsklinikum Giessen und Marburg, Giessen, Hesse
  - Klinikum der Stadt Köln gGmbH - Krankenhaus Merheim, Cologne, North Rhine-Westphalia
  - Sana-Klinikum Remscheid|Kardio, Angio, Pneumo u. Intensivmed, Remscheid, North Rhine-Westphalia
  - Charité - Universitätsmedizin Berlin, Berlin

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.